CLINICAL TRIAL: NCT03432403
Title: The Effect of Esophagogastroduodenoscopy Scope Insertion on the Intracuff Pressure of a New, Modified Laryngeal Mask Airway in Children
Brief Title: The Effect of EGD Scope Insertion on the Intracuff Pressure of a New, Modified LMA in Children
Status: Completed | Type: Observational
Sponsor: Jason Bryant (Other)
Responsible Party: Sponsor-Investigator, Jason Bryant, Anesthesiologist, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Other Study IDs: IRB17-00680
Record Dates: First submitted 2018-01-23; First posted 2018-02-14 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Intracuff Pressure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- New LMA or Old LMA: newly designed LMA or older designed LMA
  Interventions: Device: Ambu LMA; Device: Gastro LMA

INTERVENTIONS:
Device: Ambu LMA — Will be randomized to either the new Gastro LMA or old Ambu LMA for EGD procedure and the intracuff pressure will be measured
  Other Names: old LMA
Device: Gastro LMA — Will be randomized to either the new Gastro LMA or old Ambu LMA for EGD procedure and the intracuff pressure will be measured
  Other Names: new LMA

SUMMARY:
The purpose of this current study is to compare changes of the intracuff pressure in the newly designed LMA with the older design LMA after insertion of an esophagogastroduodenoscopy (EGD) probe in pediatric patients and adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Patients who weigh more than 30 kg
* Patients undergoing an EGD
* Patients getting an LMA

Exclusion Criteria:

* Patients who weigh less than 30 kg
* Use of an EGD probe with an OD greater than 14 mm
* Decision not to use an LMA for the procedure
* Tracheomalacia, bronchomalacia, or any other airway issues

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who weigh more than 30 kg who are undergoing an EGD and who are getting an LMA at Nationwide Children's Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2017-11-15 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Excessive intracuff pressure | as long as the LMA is in place in the OR with usually a max amount of time of 45 minutes
  Our primary goal is to compare the incidence of excessive intracuff pressure after EGD probe insertion between the newly designed LMA and the older version LMA. For this primary outcome, we will define excessive intracuff pressure as ≥40 cmH2O.

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States